CLINICAL TRIAL: NCT00943722
Title: A Phase III Clinical Trial to Study the Immunogenicity, Tolerability, and Manufacturing Consistency of V503 (A Multivalent Human Papillomavirus [HPV] L1 Virus-Like Particle [VLP] Vaccine) in Preadolescents and Adolescents (9 to 15 Year Olds) With a Comparison to Young Women (16 to 26 Year Olds)
Brief Title: A Study of V503 (A Multivalent Human Papillomavirus [HPV] L1 Virus-Like Particle [VLP] Vaccine) in Preadolescents and Adolescents (V503-002)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V503-002; 2009_611 (Other: Merck); 2009-011617-25 (EudraCT Number)
Record Dates: First submitted 2009-07-21; First posted 2009-07-22 (Estimated); Results first posted 2015-01-13 (Estimated); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Cervical Cancers; Vulvar Cancer; Vaginal Cancer; Genital Lesions; PAP Test Abnormalities; HPV Infections
MeSH Terms: conditions — Uterine Cervical Neoplasms; Vulvar Neoplasms; Vaginal Neoplasms; Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 9- to 15-Year-Old Females (Lot 1) (Experimental): 9-valent human papillomavirus (9vHPV) L1 VLP vaccine, 0.5 mL intramuscular injection at Day 1, Month 2, and Month 6. Vaccine dose administered is obtained from manufacturing Lot 1.
  Interventions: Biological: V503
- 9- to 15-Year-Old Females (Lot 2) (Experimental): 9-valent human papillomavirus (9vHPV) L1 VLP vaccine, 0.5 mL intramuscular injection at Day 1, Month 2, and Month 6. Vaccine dose administered is obtained from manufacturing Lot 2.
  Interventions: Biological: V503
- 9- to 15-Year-Old Females (Lot 3) (Experimental): 9-valent human papillomavirus (9vHPV) L1 VLP vaccine, 0.5 mL intramuscular injection at Day 1, Month 2, and Month 6. Vaccine dose administered is obtained from manufacturing Lot 3.
  Interventions: Biological: V503
- 9- to 15-Year-Old Males (Lot 1) (Experimental): 9-valent human papillomavirus (9vHPV) L1 VLP vaccine, 0.5 mL intramuscular injection at Day 1, Month 2, and Month 6. Vaccine dose administered is obtained from manufacturing Lot 1.
  Interventions: Biological: V503
- 16- to 26-Year-Old Females (Lot 1) (Experimental): 9-valent human papillomavirus (9vHPV) L1 VLP vaccine, 0.5 mL intramuscular injection at Day 1, Month 2, and Month 6. Vaccine dose administered is obtained from manufacturing Lot 1.
  Interventions: Biological: V503

INTERVENTIONS:
Biological: V503 — Multivalent HPV L1 VLP vaccine, 0.5 mL intramuscular injection at Day 1, Month 2, and Month 6. Vaccine dose administered is obtained from manufacturing Lots 1, 2, or 3.

SUMMARY:
This study will evaluate the immunogenicity and tolerability of V503 (a multivalent human papillomavirus [HPV] L1 virus-like particle [VLP] vaccine) in preadolescent and adolescent participants between 9 and 15 years old and demonstrate the consistency of the manufactured vaccine through assessment of 3 different final manufacturing process lots of V503.

The primary hypotheses are as follows:

1. The 9-valent HPV L1 VLP vaccine when administered to preadolescent and adolescent boys and girls 9 to 15 years of age and young women 16 to 26 years of age is generally well-tolerated.
2. 9-valent HPV L1 VLP vaccine induces non-inferior immune responses in preadolescent and adolescent girls 9 to 15 years of age who are seronegative at Day 1 to the relevant HPV type compared to young women 16 to 26 years of age who are seronegative at Day 1 and polymerase chain reaction (PCR)-negative Day 1 through Month 7 to the relevant HPV type, as measured by anti-HPV 6, 11, 16, 18, 31, 33, 45, 52, and 58 geometric mean titers (GMTs) at 4 weeks post-dose 3.
3. The 9-valent HPV L1 VLP vaccine induces non-inferior immune responses in preadolescent and adolescent boys 9 to 15 years of age who are seronegative at Day 1 to the relevant HPV type compared to young women 16 to 26 years of age who are seronegative at Day 1 and PCR-negative Day 1 through Month 7 to the relevant HPV type, as measured by anti-HPV 6, 11, 16, 18, 31, 33, 45, 52, and 58 GMTs at 4 weeks post-dose 3.
4. Three separate final manufacturing process (FMP) lots of the 9-valent HPV L1 VLP vaccine induce similar immune responses, as measured by anti-HPV types 6, 11, 16, 18, 31, 33, 45, 52, and 58 GMTs at 4 weeks post-dose 3.

DETAILED DESCRIPTION:
The base study V503-002 was a 12-month study that collected immunogenicity data through Month 7 and safety data through Month 12.

An optional extension study (V503-002 EXT1) collected safety and immunogenicity information through Month 36. Participants enrolled in the 16- to 26-year-old cohort in the base study were not included in EXT1. Per protocol, EXT1 included immunogenicity data from a subset of 9- to 15-year-old females and safety data from all 9- to 15-year-old females regardless of lot administered.

An optional second extension study (V503-002 EXT2) collected long-term safety and immunogenicity information through approximately Month 126. No study vaccine was administered in the extension studies. Participants enrolled in the 16- to 26-year-old cohort in the base study were not included in EXT2. Per protocol, EXT2 included immunogenicity data from a subset of 9- to 15-year-old females and effectiveness and safety data from all 9- to 15-year-old females regardless of lot administered.

ELIGIBILITY:
Inclusion Criteria:

Boys and Girls Age 9 to 15:

* Participant has not had sexual intercourse prior to the study and does not plan to become sexually active during the study period Day 1 to Month 7

Women Age 16 to 26:

* Participant has never had Pap testing or has had only normal results
* Participant has had 0 to 4 sexual partners at the time of enrollment

Exclusion Criteria:

Boys and Girls Age 9 to 15:

* History of allergic reaction that required medical intervention
* Currently enrolled in any other clinical study
* Participant is pregnant
* Participant is immunocompromised or has taken immunosuppressants in the last year
* Participant has received a marketed HPV vaccine or participated in an HPV vaccine clinical trial
* Participant has a history of positive test for HPV

Women Age 16 to 26:

* History of allergic reaction that required medical intervention
* Currently enrolled in any other clinical study
* Participant is pregnant
* Participant is immunocompromised or has taken immunosuppressants in the last year
* Participant has received a marketed HPV vaccine or participated in an HPV vaccine clinical trial
* Participant has a history of positive test for HPV
* Participant has a history of abnormal cervical biopsy result
* Participant has a history of external genital lesions

Ages: 9 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3074 (Actual)
Dates: Start 2009-08-27 (Actual); Primary Completion 2011-04-30 (Actual); Study Completion 2021-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Luxembourg A, Moreira ED Jr, Samakoses R, Kim KH, Sun X, Maansson R, Moeller E, Christiano S, Chen J. Phase III, randomized controlled trial in girls 9-15 years old to evaluate lot consistency of a novel nine-valent human papillomavirus L1 virus-like particle vaccine. Hum Vaccin Immunother. 2015;11(6):1306-12. doi: 10.1080/21645515.2015.1009819. PMID 26086587
- [Result] Van Damme P, Olsson SE, Block S, Castellsague X, Gray GE, Herrera T, Huang LM, Kim DS, Pitisuttithum P, Chen J, Christiano S, Maansson R, Moeller E, Sun X, Vuocolo S, Luxembourg A. Immunogenicity and Safety of a 9-Valent HPV Vaccine. Pediatrics. 2015 Jul;136(1):e28-39. doi: 10.1542/peds.2014-3745. PMID 26101366
- [Result] Moreira ED Jr, Block SL, Ferris D, Giuliano AR, Iversen OE, Joura EA, Kosalaraksa P, Schilling A, Van Damme P, Bornstein J, Bosch FX, Pils S, Cuzick J, Garland SM, Huh W, Kjaer SK, Qi H, Hyatt D, Martin J, Moeller E, Ritter M, Baudin M, Luxembourg A. Safety Profile of the 9-Valent HPV Vaccine: A Combined Analysis of 7 Phase III Clinical Trials. Pediatrics. 2016 Aug;138(2):e20154387. doi: 10.1542/peds.2015-4387. Epub 2016 Jul 15. PMID 27422279
- [Result] Olsson SE, Restrepo JA, Reina JC, Pitisuttithum P, Ulied A, Varman M, Van Damme P, Moreira ED Jr, Ferris D, Block S, Bautista O, Gallagher N, McCauley J, Luxembourg A. Long-term immunogenicity, effectiveness, and safety of nine-valent human papillomavirus vaccine in girls and boys 9 to 15 years of age: Interim analysis after 8 years of follow-up. Papillomavirus Res. 2020 Dec;10:100203. doi: 10.1016/j.pvr.2020.100203. Epub 2020 Jul 11. PMID 32659510
- [Derived] Restrepo J, Herrera T, Samakoses R, Reina JC, Pitisuttithum P, Ulied A, Bekker LG, Moreira ED, Olsson SE, Block SL, Hammes LS, Laginha F, Ferenczy A, Kurman R, Ronnett BM, Stoler M, Bautista O, Gallagher NE, Salituro G, Ye M, Luxembourg A. Ten-Year Follow-up of 9-Valent Human Papillomavirus Vaccine: Immunogenicity, Effectiveness, and Safety. Pediatrics. 2023 Oct 1;152(4):e2022060993. doi: 10.1542/peds.2022-060993. PMID 37667847
- [Derived] Garland SM, Pitisuttithum P, Ngan HYS, Cho CH, Lee CY, Chen CA, Yang YC, Chu TY, Twu NF, Samakoses R, Takeuchi Y, Cheung TH, Kim SC, Huang LM, Kim BG, Kim YT, Kim KH, Song YS, Lalwani S, Kang JH, Sakamoto M, Ryu HS, Bhatla N, Yoshikawa H, Ellison MC, Han SR, Moeller E, Murata S, Ritter M, Sawata M, Shields C, Walia A, Perez G, Luxembourg A. Efficacy, Immunogenicity, and Safety of a 9-Valent Human Papillomavirus Vaccine: Subgroup Analysis of Participants From Asian Countries. J Infect Dis. 2018 Jun 5;218(1):95-108. doi: 10.1093/infdis/jiy133. PMID 29767739
- [Derived] Ruiz-Sternberg AM, Moreira ED Jr, Restrepo JA, Lazcano-Ponce E, Cabello R, Silva A, Andrade R, Revollo F, Uscanga S, Victoria A, Guevara AM, Luna J, Plata M, Dominguez CN, Fedrizzi E, Suarez E, Reina JC, Ellison MC, Moeller E, Ritter M, Shields C, Cashat M, Perez G, Luxembourg A. Efficacy, immunogenicity, and safety of a 9-valent human papillomavirus vaccine in Latin American girls, boys, and young women. Papillomavirus Res. 2018 Jun;5:63-74. doi: 10.1016/j.pvr.2017.12.004. Epub 2017 Dec 19. PMID 29269325

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The base study was a 12-month study that collected immunogenicity data through Month 7 and safety data through Month 12.
Pre-assignment Details: Extension study 1 (EXT1) collected data to Month 36. Extension study 2 (EXT2) collected long-term data through ~Month 126. No study vaccine was administered.
  Per protocol, participants enrolled in the 16- to 26-year-old arm in the base study were not included in the extension study.
  Per protocol, the extension study included data from 9- to 15-year-old females regardless of lot administered (arm: "Extension Study: 9- to 15- Year Old Females").
Groups:
- Base Study: 9- to 15-Year-Old Females (Lot 1): 9-valent human papillomavirus (9vHPV) L1 virus-like particle (VLP) vaccine, 0.5 mL intramuscular injection at Day 1, Month 2, and Month 6. Vaccine dose administered was obtained from manufacturing Lot 1.
- Base Study: 9- to 15-Year-Old Females (Lot 2): 9vHPV L1 VLP vaccine, 0.5 mL intramuscular injection at Day 1, Month 2, and Month 6. Vaccine dose administered was obtained from manufacturing Lot 2.
- Base Study: 9- to 15-Year-Old Females (Lot 3): 9vHPV L1 VLP vaccine, 0.5 mL intramuscular injection at Day 1, Month 2, and Month 6. Vaccine dose administered was obtained from manufacturing Lot 3.
- Base Study: 9- to 15-Year-Old Males (Lot 1); Base Study: 16- to 26-Year-Old Females (Lot 1): 9vHPV L1 VLP vaccine, 0.5 mL intramuscular injection at Day 1, Month 2, and Month 6. Vaccine dose administered was obtained from manufacturing Lot 1.
- Extension Study: 9- to 15-Year-Old Females; Extension Study: 9- to 15-Year-Old Males: In the base study, participants received the 9vHPV L1 VLP vaccine (0.5 mL intramuscular injection) at Day 1, Month 2, and Month 6 and were evaluated through Month 12. In the extension studies, the participants were followed up for safety and immunogenicity up to Month 36 (EXT1) and for immunogenicity, effectiveness, and safety up to Month 126 (EXT2).
Period: Base Study
Arm/Group | Base Study: 9- to 15-Year-Old Females (Lot 1) | Base Study: 9- to 15-Year-Old Females (Lot 2) | Base Study: 9- to 15-Year-Old Females (Lot 3) | Base Study: 9- to 15-Year-Old Males (Lot 1) | Base Study: 16- to 26-Year-Old Females (Lot 1) | Extension Study: 9- to 15-Year-Old Females | Extension Study: 9- to 15-Year-Old Males
Started | 648 | 643 | 644 | 669 | 470 | 0 | 0
Vaccination 1 | 646 | 642 | 644 | 666 | 468 | 0 | 0
Vaccination 2 | 637 | 633 | 638 | 658 | 462 | 0 | 0
Vaccination 3 | 635 | 627 | 637 | 653 | 455 | 0 | 0
At Least One Dose With Protocol-specified Safety Follow-up | 643 | 639 | 641 | 662 | 466 | 0 | 0
Completed | 623 | 621 | 631 | 647 | 444 | 0 | 0
Not Completed | 25 | 22 | 13 | 22 | 26 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 12 | 8 | 10 | 8 | 11 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 1 | 0 | 2 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 12 | 13 | 2 | 13 | 8 | 0 | 0
Not completed — Month 12 visit not completed | 0 | 0 | 0 | 0 | 2 | 0 | 0
Period: First Extension Study: EXT 1
Arm/Group | Base Study: 9- to 15-Year-Old Females (Lot 1) | Base Study: 9- to 15-Year-Old Females (Lot 2) | Base Study: 9- to 15-Year-Old Females (Lot 3) | Base Study: 9- to 15-Year-Old Males (Lot 1) | Base Study: 16- to 26-Year-Old Females (Lot 1) | Extension Study: 9- to 15-Year-Old Females | Extension Study: 9- to 15-Year-Old Males
Started (The optional EXT1 included eligible participants from the base study, with the exception of 16-26 year old females.) | 0 | 0 | 0 | 0 | 0 | 1604 | 568
Completed | 0 | 0 | 0 | 0 | 0 | 1489 | 527
Not Completed | 0 | 0 | 0 | 0 | 0 | 115 | 41
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 38 | 10
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 32 | 10
Not completed — Disposition Unknown | 0 | 0 | 0 | 0 | 0 | 44 | 21
Period: Second Extension Study: EXT 2
Arm/Group | Base Study: 9- to 15-Year-Old Females (Lot 1) | Base Study: 9- to 15-Year-Old Females (Lot 2) | Base Study: 9- to 15-Year-Old Females (Lot 3) | Base Study: 9- to 15-Year-Old Males (Lot 1) | Base Study: 16- to 26-Year-Old Females (Lot 1) | Extension Study: 9- to 15-Year-Old Females | Extension Study: 9- to 15-Year-Old Males
Started (The optional EXT2 included eligible participants from the base study, with the exception of 16-26 year old females.) | 0 | 0 | 0 | 0 | 0 | 971 | 301
Completed | 0 | 0 | 0 | 0 | 0 | 720 | 202
Not Completed | 0 | 0 | 0 | 0 | 0 | 251 | 99
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 111 | 46
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 3
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 137 | 50

BASELINE CHARACTERISTICS:
Population: Per protocol, baseline characteristics were analyzed in all participants randomized in the base study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Base Study: 9- to 15-Year-Old Females (Lot 1) | Base Study: 9- to 15-Year-Old Females (Lot 2) | Base Study: 9- to 15-Year-Old Females (Lot 3) | Base Study: 9- to 15-Year-Old Males (Lot 1) | Base Study: 16- to 26-Year-Old Females (Lot 1) | Total
Number analyzed (Participants) | 648 | 643 | 644 | 669 | 470 | 3074
Age, Customized [Number; unit: Participants]
  9 to 12 years | 440 | 432 | 432 | 450 | 0 | 1754
  13 to 15 years | 208 | 211 | 212 | 219 | 0 | 850
  16 to 26 years | 0 | 0 | 0 | 0 | 470 | 470
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 648 | 643 | 644 | 0 | 470 | 2405
  Male | 0 | 0 | 0 | 669 | 0 | 669

OUTCOME MEASURES:

1. Primary Outcome: Base Study: Geometric Mean Titers (GMTs) for Each of the HPV Types Contained in the Vaccine (9- to 15-Year-Old Females [Lot 1] and 16- to 26-Year-Old Females [Lot 1])
Description: Serum antibody titers for HPV virus-like particles (VLPs), Types 6, 11, 16, 18, 31, 33, 45, 52 and 58 were determined 4 weeks post-vaccination 3 using a competitive luminex immunoassay (cLIA). Titers were reported in milli Merck Units/mL.
Time Frame: 4 weeks post-vaccination 3 (Month 7)
Population: 9-15-year-old females and 16-26-year-old females who received 3 vaccinations from Lot 1 and met following criteria for at least 1 of the 9 HPV types: no general protocol violations, received all 3 vaccinations within acceptable day ranges, seronegative at Day 1 for HPV type(s), and had a Month 7 serum sample collected within an acceptable day range.
Measure: Geometric Mean (95% Confidence Interval); unit: milli Merck Units/mL
Arm/Group | Base Study: 9- to 15-Year-Old Females (Lot 1) | Base Study: 9- to 15-Year-Old Males (Lot 1)
Number analyzed (Participants) | 535 | 378
milli Merck Units/mL
  Anti-HPV 6: number analyzed (Participants) | 517 | 328
  Anti-HPV 6 | 1715.4 [1595.1 to 1844.7] | 900.8 [822.3 to 986.9]
  Anti-HPV 11: number analyzed (Participants) | 517 | 332
  Anti-HPV 11 | 1295.1 [1204.1 to 1393.0] | 706.6 [645.2 to 773.8]
  Anti-HPV 16: number analyzed (Participants) | 529 | 329
  Anti-HPV 16 | 6979.8 [6508.1 to 7485.8] | 3522.6 [3223.5 to 3849.5]
  Anti-HPV 18: number analyzed (Participants) | 531 | 345
  Anti-HPV 18 | 2153.7 [1980.4 to 2342.1] | 882.7 [795.4 to 979.5]
  Anti-HPV 31: number analyzed (Participants) | 522 | 340
  Anti-HPV 31 | 1891.6 [1745.7 to 2049.7] | 753.9 [682.5 to 832.7]
  Anti-HPV 33: number analyzed (Participants) | 534 | 354
  Anti-HPV 33 | 980.4 [911.7 to 1054.3] | 466.8 [426.9 to 510.3]
  Anti-HPV 45: number analyzed (Participants) | 534 | 368
  Anti-HPV 45 | 714.4 [651.9 to 782.8] | 272.2 [243.8 to 303.9]
  Anti-HPV 52: number analyzed (Participants) | 533 | 337
  Anti-HPV 52 | 932.9 [864.8 to 1006.4] | 419.6 [381.4 to 461.5]
  Anti-HPV 58: number analyzed (Participants) | 531 | 332
  Anti-HPV 58 | 1286.7 [1195.7 to 1384.6] | 590.5 [538.2 to 647.9]
Statistical Analysis 1: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Males (Lot 1); Anti-HPV 6; Test type: Non-Inferiority — non-inferiority requires that the lower bound of two-sided 95% confidence interval (CI) of GMT ratio be greater than 0.67; p < 0.001, ANOVA — one-sided tests of non-inferiority conducted at the alpha=0.025 level; model with a response of log individual titers and a fixed effect for comparison group; model with a response of log individual titers and a fixed effect for comparison group; GMT ratio = 1.90, 95% CI 2-sided [1.70 to 2.14] — GMT ratio = GMT for 9- to 15-Year-Old Females (Lot 1) divided by GMT for 16- to 26-Year-Old Females (Lot 1)
Statistical Analysis 2: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Males (Lot 1); Anti-HPV 11; Test type: Non-Inferiority — Non-inferiority requires that the lower bound of two-sided 95% CI of GMT ratio be greater than 0.67; p < 0.001, ANOVA — [p-value comment as in outcome 1, analysis 1]; model with a response of log individual titers and a fixed effect for comparison group; GMT ratio = 1.83, 95% CI 2-sided [1.63 to 2.06] — GMT ratio = GMT for 9- to 15-Year-Old Females (Lot 1) divided by GMT for 16- to 26-Year-Old Females (Lot 1)
Statistical Analysis 3: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Males (Lot 1); Anti-HPV 16; Test type: Non-Inferiority — Non-inferiority requires that the lower bound of two-sided 95% CI of GMT ratio be greater than 0.67; p < 0.001, ANOVA — [p-value comment as in outcome 1, analysis 1]; model with a response of log individual titers and a fixed effect for comparison group; GMT ratio = 1.98, 95% CI 2-sided [1.77 to 2.22] — GMT ratio = GMT for 9- to 15-Year-Old Females (Lot 1) divided by GMT for 16- to 26-Year-Old Females (Lot 1)
Statistical Analysis 4: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Males (Lot 1); Anti-HPV 18; Test type: Non-Inferiority — non-inferiority requires that the lower bound of two-sided 95% CI of GMT ratio be greater than 0.67; p < 0.001, ANOVA — [p-value comment as in outcome 1, analysis 1]; model with a response of log individual titers and a fixed effect for comparison group; GMT ratio = 2.44, 95% CI 2-sided [2.13 to 2.80] — GMT ratio = GMT for 9- to 15-Year-Old Females (Lot 1) divided by GMT for 16- to 26-Year-Old Females (Lot 1)
Statistical Analysis 5: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Males (Lot 1); Anti-HPV 31; Test type: Non-Inferiority — non-inferiority requires that the lower bound of two-sided 95% CI of GMT ratio be greater than 0.67; p < 0.001, ANOVA — [p-value comment as in outcome 1, analysis 1]; model with a response of log individual titers and a fixed effect for comparison group; GMT ratio = 2.51, 95% CI 2-sided [2.21 to 2.85] — GMT ratio = GMT for 9- to 15-Year-Old Females (Lot 1) divided by GMT for 16- to 26-Year-Old Females (Lot 1)
Statistical Analysis 6: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Males (Lot 1); Anti-HPV 33; Test type: Non-Inferiority — non-inferiority requires that the lower bound of two-sided 95% CI of GMT ratio be greater than 0.67; p < 0.001, ANOVA — [p-value comment as in outcome 1, analysis 1]; model with a response of log individual titers and a fixed effect for comparison group; GMT ratio = 2.10, 95% CI 2-sided [1.87 to 2.36] — GMT ratio = GMT for 9- to 15-Year-Old Females (Lot 1) divided by GMT for 16- to 26-Year-Old Females (Lot 1)
Statistical Analysis 7: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Males (Lot 1); Anti-HPV 45; Test type: Non-Inferiority — non-inferiority requires that the lower bound of two-sided 95% CI of GMT ratio be greater than 0.67; p < 0.001, ANOVA — [p-value comment as in outcome 1, analysis 1]; model with a response of log individual titers and a fixed effect for comparison group; GMT ratio = 2.62, 95% CI 2-sided [2.27 to 3.03] — GMT ratio = GMT for 9- to 15-Year-Old Females (Lot 1) divided by GMT for 16- to 26-Year-Old Females (Lot 1)
Statistical Analysis 8: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Males (Lot 1); Anti-HPV 52; Test type: Non-Inferiority — non-inferiority requires that the lower bound of two-sided 95% CI of GMT ratio be greater than 0.67; p < 0.001, ANOVA — [p-value comment as in outcome 1, analysis 1]; model with a response of log individual titers and a fixed effect for comparison group; GMT ratio = 2.22, 95% CI 2-sided [1.97 to 2.51] — GMT ratio = GMT for 9- to 15-Year-Old Females (Lot 1) divided by GMT for 16- to 26-Year-Old Females (Lot 1)
Statistical Analysis 9: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Males (Lot 1); Anti-HPV 58; Test type: Non-Inferiority — non-inferiority requires that the lower bound of two-sided 95% CI of GMT ratio be greater than 0.67; p < 0.001, ANOVA — [p-value comment as in outcome 1, analysis 1]; model with a response of log individual titers and a fixed effect for comparison group; GMT ratio = 2.18, 95% CI 2-sided [1.93 to 2.45] — GMT ratio = GMT for 9- to 15-Year-Old Females (Lot 1) divided by GMT for 16- to 26-Year-Old Females (Lot 1)

2. Primary Outcome: Base Study: GMTs for Each of the HPV Types Contained in the Vaccine (9- to 15-Year-Old Males [Lot 1] and 16- to 26-Year-Old Females [Lot 1])
Description: Serum antibody titers for HPV VLPs, Types 6, 11, 16, 18, 31, 33, 45, 52 and 58 were determined 4 weeks post-vaccination 3 using a competitive luminex immunoassay (cLIA). Titers were reported in milli Merck Units/mL.
Time Frame: 4 weeks post-vaccination 3 (Month 7)
Population: 9-15-year-old males and 16-26-year-old females who received 3 vaccinations from Lot 1 and met following criteria for at least 1 of the 9 HPV types: no general protocol violations, received all 3 vaccinations within acceptable day ranges, seronegative at Day 1 for HPV type(s), and had a Month 7 serum sample collected within an acceptable day range.
Measure: Geometric Mean (95% Confidence Interval); unit: milli Merck Units/mL
Arm/Group | Base Study: 9- to 15-Year-Old Males (Lot 1) | Base Study: 16- to 26-Year-Old Females (Lot 1)
Number analyzed (Participants) | 570 | 378
milli Merck Units/mL
  Anti-HPV 6: number analyzed (Participants) | 559 | 328
  Anti-HPV 6 | 2084.7 [1944.0 to 2235.7] | 900.8 [822.3 to 986.9]
  Anti-HPV 11: number analyzed (Participants) | 559 | 332
  Anti-HPV 11 | 1487.1 [1386.5 to 1595.0] | 706.6 [645.2 to 773.8]
  Anti-HPV 16: number analyzed (Participants) | 569 | 329
  Anti-HPV 16 | 8628.9 [8065.9 to 9231.3] | 3522.6 [3223.5 to 3849.5]
  Anti-HPV 18: number analyzed (Participants) | 567 | 345
  Anti-HPV 18 | 2822.8 [2602.8 to 3061.5] | 882.7 [795.4 to 979.5]
  Anti-HPV 31: number analyzed (Participants) | 564 | 340
  Anti-HPV 31 | 2221.2 [2056.1 to 2399.5] | 753.9 [682.5 to 832.7]
  Anti-HPV 33: number analyzed (Participants) | 567 | 354
  Anti-HPV 33 | 1198.7 [1117.1 to 1286.2] | 466.8 [426.9 to 510.3]
  Anti-HPV 45: number analyzed (Participants) | 570 | 368
  Anti-HPV 45 | 907.0 [830.2 to 991.0] | 272.2 [243.8 to 303.9]
  Anti-HPV 52: number analyzed (Participants) | 568 | 337
  Anti-HPV 52 | 1037.8 [964.4 to 1116.9] | 419.6 [381.4 to 461.5]
  Anti-HPV 58: number analyzed (Participants) | 566 | 332
  Anti-HPV 58 | 1567.7 [1460.2 to 1683.1] | 590.5 [538.2 to 647.9]
Statistical Analysis 1: Comparison: Base Study: 9- to 15-Year-Old Males (Lot 1) vs Base Study: 16- to 26-Year-Old Females (Lot 1); Anti-HPV 6; Test type: Non-Inferiority — non-inferiority requires that the lower bound of two-sided 95% CI of GMT ratio be greater than 0.67; p < 0.001, ANOVA — [p-value comment as in outcome 1, analysis 1]; model with a response of log individual titers and a fixed effect for comparison group; GMT ratio = 2.31, 95% CI 2-sided [2.07 to 2.59] — GMT ratio = GMT for 9- to 15-Year-Old males (Lot 1) divided by GMT for 16- to 26-Year-Old Females (Lot 1)
Statistical Analysis 2: Comparison: Base Study: 9- to 15-Year-Old Males (Lot 1) vs Base Study: 16- to 26-Year-Old Females (Lot 1); Anti-HPV 11; Test type: Non-Inferiority — non-inferiority requires that the lower bound of two-sided 95% CI of GMT ratio be greater than 0.67; p < 0.001, ANOVA — [p-value comment as in outcome 1, analysis 1]; model with a response of log individual titers and a fixed effect for comparison group; GMT ratio = 2.10, 95% CI 2-sided [1.88 to 2.36] — GMT ratio = GMT for 9- to 15-Year-Old Males (Lot 1) divided by GMT for 16- to 26-Year-Old Females (Lot 1)
Statistical Analysis 3: Comparison: Base Study: 9- to 15-Year-Old Males (Lot 1) vs Base Study: 16- to 26-Year-Old Females (Lot 1); Anti-HPV 16; Test type: Non-Inferiority — non-inferiority requires that the lower bound of two-sided 95% CI of GMT ratio be greater than 0.67; p < 0.001, ANOVA — [p-value comment as in outcome 1, analysis 1]; model with a response of log individual titers and a fixed effect for comparison group; GMT ratio = 2.45, 95% CI 2-sided [2.19 to 2.74] — GMT ratio = GMT for 9- to 15-Year-Old Males (Lot 1) divided by GMT for 16- to 26-Year-Old Females (Lot 1)
Statistical Analysis 4: Comparison: Base Study: 9- to 15-Year-Old Males (Lot 1) vs Base Study: 16- to 26-Year-Old Females (Lot 1); Anti-HPV 18; Test type: Non-Inferiority — non-inferiority requires that the lower bound of two-sided 95% CI of GMT ratio be greater than 0.67; p < 0.001, ANOVA — [p-value comment as in outcome 1, analysis 1]; model with a response of log individual titers and a fixed effect for comparison group; GMT ratio = 3.20, 95% CI 2-sided [2.80 to 3.65] — GMT ratio = GMT for 9- to 15-Year-Old Males (Lot 1) divided by GMT for 16- to 26-Year-Old Females (Lot 1)
Statistical Analysis 5: Comparison: Base Study: 9- to 15-Year-Old Males (Lot 1) vs Base Study: 16- to 26-Year-Old Females (Lot 1); Anti-HPV 31; Test type: Non-Inferiority — non-inferiority requires that the lower bound of two-sided 95% CI of GMT ratio be greater than 0.67; p < 0.001, ANOVA — [p-value comment as in outcome 1, analysis 1]; model with a response of log individual titers and a fixed effect for comparison group; GMT ratio = 2.95, 95% CI 2-sided [2.60 to 3.34] — GMT ratio = GMT for 9- to 15-Year-Old Males (Lot 1) divided by GMT for 16- to 26-Year-Old Females (Lot 1)
Statistical Analysis 6: Comparison: Base Study: 9- to 15-Year-Old Males (Lot 1) vs Base Study: 16- to 26-Year-Old Females (Lot 1); Anti-HPV 33; Test type: Non-Inferiority — non-inferiority requires that the lower bound of two-sided 95% CI of GMT ratio be greater than 0.67; p < 0.001, ANOVA — [p-value comment as in outcome 1, analysis 1]; model with a response of log individual titers and a fixed effect for comparison group; GMT ratio = 2.57, 95% CI 2-sided [2.29 to 2.88] — GMT ratio = GMT for 9- to 15-Year-Old Males (Lot 1) divided by GMT for 16- to 26-Year-Old Females (Lot 1)
Statistical Analysis 7: Comparison: Base Study: 9- to 15-Year-Old Males (Lot 1) vs Base Study: 16- to 26-Year-Old Females (Lot 1); Anti-HPV 45; Test type: Non-Inferiority — non-inferiority requires that the lower bound of two-sided 95% CI of GMT ratio be greater than 0.67; p < 0.001, ANOVA — [p-value comment as in outcome 1, analysis 1]; model with a response of log individual titers and a fixed effect for comparison group; GMT ratio = 3.33, 95% CI 2-sided [2.89 to 3.84] — GMT ratio = GMT for 9- to 15-Year-Old Males (Lot 1) divided by GMT for 16- to 26-Year-Old Females (Lot 1)
Statistical Analysis 8: Comparison: Base Study: 9- to 15-Year-Old Males (Lot 1) vs Base Study: 16- to 26-Year-Old Females (Lot 1); Anti-HPV 52; Test type: Non-Inferiority — non-inferiority requires that the lower bound of two-sided 95% CI of GMT ratio be greater than 0.67; p < 0.001, ANOVA — [p-value comment as in outcome 1, analysis 1]; model with a response of log individual titers and a fixed effect for comparison group; GMT ratio = 2.47, 95% CI 2-sided [2.19 to 2.79] — GMT ratio = GMT for 9- to 15-Year-Old Males (Lot 1) divided by GMT for 16- to 26-Year-Old Females (Lot 1)
Statistical Analysis 9: Comparison: Base Study: 9- to 15-Year-Old Males (Lot 1) vs Base Study: 16- to 26-Year-Old Females (Lot 1); Anti-HPV 58; Test type: Non-Inferiority — non-inferiority requires that the lower bound of two-sided 95% CI of GMT ratio be greater than 0.67; p < 0.001, ANOVA — [p-value comment as in outcome 1, analysis 1]; model with a response of log individual titers and a fixed effect for comparison group; GMT ratio = 2.66, 95% CI 2-sided [2.37 to 2.98] — GMT ratio = GMT for 9- to 15-Year-Old Males (Lot 1) divided by GMT for 16- to 26-Year-Old Females (Lot 1)

3. Primary Outcome: Base Study: GMTs for Each of the HPV Types Contained in the Vaccine (Lot Consistency Study)
Description: Serum antibody titers for HPV VLPs, Types 6, 11, 16, 18, 31, 33, 45, 52 and 58 were determined 4 weeks post-vaccination 3 using cLIA. Titers were reported in milli Merck Units/mL.
Time Frame: 4 weeks post-vaccination 3 (Month 7)
Population: 9-15-year-old females who received 3 vaccinations from Lots 1, 2, or 3 and met following criteria for at least 1 of the 9 HPV types: no general protocol violations, received all 3 vaccinations within acceptable day ranges, seronegative at Day 1 for HPV type(s), and had a Month 7 serum sample collected within an acceptable day range.
Measure: Geometric Mean (95% Confidence Interval); unit: milli Merck Units/mL
Arm/Group | Base Study: 9- to 15-Year-Old Females (Lot 1) | Base Study: 9- to 15-Year-Old Females (Lot 2) | Base Study: 9- to 15-Year-Old Females (Lot 3)
Number analyzed (Participants) | 535 | 549 | 565
milli Merck Units/mL
  Anti-HPV 6: number analyzed (Participants) | 517 | 536 | 544
  Anti-HPV 6 | 1715.4 [1588.7 to 1852.2] | 1763.3 [1635.4 to 1901.3] | 1659.9 [1540.3 to 1788.7]
  Anti-HPV 11: number analyzed (Participants) | 517 | 536 | 544
  Anti-HPV 11 | 1295.1 [1197.8 to 1400.3] | 1311.7 [1214.9 to 1416.3] | 1232.0 [1141.7 to 1329.5]
  Anti-HPV 16: number analyzed (Participants) | 529 | 542 | 556
  Anti-HPV 16 | 6979.8 [6476.1 to 7522.8] | 7292.9 [6772.7 to 7853.1] | 6948.2 [6458.7 to 7474.9]
  Anti-HPV 18: number analyzed (Participants) | 531 | 547 | 563
  Anti-HPV 18 | 2153.7 [1970.9 to 2353.5] | 2134.1 [1955.6 to 2329.0] | 1966.6 [1804.3 to 2143.5]
  Anti-HPV 31: number analyzed (Participants) | 522 | 542 | 553
  Anti-HPV 31 | 1891.6 [1738.5 to 2058.2] | 1867.8 [1719.3 to 2029.1] | 1879.0 [1731.0 to 2039.6]
  Anti-HPV 33: number analyzed (Participants) | 534 | 543 | 560
  Anti-HPV 33 | 980.4 [909.2 to 1057.2] | 922.7 [856.2 to 994.4] | 931.1 [865.0 to 1002.3]
  Anti-HPV 45: number analyzed (Participants) | 534 | 548 | 565
  Anti-HPV 45 | 714.4 [650.1 to 785.0] | 827.7 [754.1 to 908.5] | 678.4 [619.0 to 743.6]
  Anti-HPV 52: number analyzed (Participants) | 533 | 547 | 562
  Anti-HPV 52 | 932.9 [860.8 to 1011.0] | 1007.9 [931.0 to 1091.2] | 971.2 [898.1 to 1050.3]
  Anti-HPV 58: number analyzed (Participants) | 531 | 539 | 560
  Anti-HPV 58 | 1286.7 [1190.0 to 1391.3] | 1344.9 [1244.6 to 1453.3] | 1208.1 [1119.6 to 1303.6]
Statistical Analysis 1: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Females (Lot 2); Anti-HPV 6; Test type: Equivalence — equivalence requires that the two-sided 95% CI for the ratio of the GMTs be entirely contained within the interval (0.5, 2.0); GMT ratio = 0.97, 95% CI 2-sided [0.88 to 1.08] — GMT ratio = GMT for 9- to 15-Year-Old Females (Lot 1) divided by GMT for 9- to 15-Year-Old Females (Lot 2)
Statistical Analysis 2: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Females (Lot 3); Anti-HPV 6; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; GMT ratio = 1.03, 95% CI 2-sided [0.93 to 1.16] — GMT ratio = GMT for 9- to 15-Year-Old Females (Lot 1) divided by GMT for 9- to 15-Year-Old Females (Lot 3)
Statistical Analysis 3: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 2) vs Base Study: 9- to 15-Year-Old Females (Lot 3); Anti-HPV 6; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; GMT ratio = 1.06, 95% CI 2-sided [0.95 to 1.19] — GMT ratio = GMT for 9- to 15-Year-Old Females (Lot 2) divided by GMT for 9- to 15-Year-Old Females (Lot 3)
Statistical Analysis 4: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Females (Lot 2); Anti-HPV 11; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; GMT ratio = 1.00, 95% CI 2-sided [0.90 to 1.11] — GMT ratio = GMT for 9- to 15-Year-Old Females (Lot 1) divided by GMT for 9- to 15-Year-Old Females (Lot 2)
Statistical Analysis 5: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Females (Lot 3); Anti-HPV 11; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; GMT ratio = 1.07, 95% CI 2-sided [0.95 to 1.20] — GMT ratio = GMT for 9- to 15-Year-Old Females (Lot 1) divided by GMT for 9- to 15-Year-Old Females (Lot 3)
Statistical Analysis 6: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 2) vs Base Study: 9- to 15-Year-Old Females (Lot 3); Anti-HPV 11; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; GMT ratio = 1.07, 95% CI 2-sided [0.95 to 1.20] — GMT ratio = GMT for 9- to 15-Year-Old Females (Lot 2) divided by GMT for 9- to 15-Year-Old Females (Lot 3)
Statistical Analysis 7: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Females (Lot 2); Anti-HPV 16; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; GMT ratio = 0.96, 95% CI 2-sided [0.86 to 1.06] — GMT ratio = GMT for 9- to 15-Year-Old Females (Lot 1) divided by GMT for 9- to 15-Year-Old Females (Lot 2)
Statistical Analysis 8: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Females (Lot 3); Anti-HPV 16; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; GMT ratio = 1.00, 95% CI 2-sided [0.90 to 1.12] — GMT ratio = GMT for 9- to 15-Year-Old Females (Lot 1) divided by GMT for 9- to 15-Year-Old Females (Lot 3)
Statistical Analysis 9: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 2) vs Base Study: 9- to 15-Year-Old Females (Lot 3); Anti-HPV 16; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; GMT ratio = 1.05, 95% CI 2-sided [0.94 to 1.17] — GMT ratio = GMT for 9- to 15-Year-Old Females (Lot 2) divided by GMT for 9- to 15-Year-Old Females (Lot 3)
Statistical Analysis 10: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Females (Lot 2); Anti-HPV 18; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; GMT ratio = 1.00, 95% CI 2-sided [0.89 to 1.14] — GMT ratio = GMT for 9- to 15-Year-Old Females (Lot 1) divided by GMT for 9- to 15-Year-Old Females (Lot 2)
Statistical Analysis 11: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Females (Lot 3); Anti-HPV 18; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; GMT ratio = 1.11, 95% CI 2-sided [0.98 to 1.26] — GMT ratio = GMT for 9- to 15-Year-Old Females (Lot 1) divided by GMT for 9- to 15-Year-Old Females (Lot 3)
Statistical Analysis 12: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 2) vs Base Study: 9- to 15-Year-Old Females (Lot 3); Anti-HPV 18; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; GMT ratio = 1.11, 95% CI 2-sided [0.97 to 1.26] — GMT ratio = GMT for 9- to 15-Year-Old Females (Lot 2) divided by GMT for 9- to 15-Year-Old Females (Lot 3)
Statistical Analysis 13: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Females (Lot 2); Anti-HPV 31; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; GMT ratio = 1.00, 95% CI 2-sided [0.89 to 1.13] — GMT ratio = GMT for 9- to 15-Year-Old Females (Lot 1) divided by GMT for 9- to 15-Year-Old Females (Lot 2)
Statistical Analysis 14: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Females (Lot 3); Anti-HPV 31; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; GMT ratio = 1.02, 95% CI 2-sided [0.91 to 1.16] — GMT ratio = GMT for 9- to 15-Year-Old Females (Lot 1) divided by GMT for 9- to 15-Year-Old Females (Lot 3)
Statistical Analysis 15: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 2) vs Base Study: 9- to 15-Year-Old Females (Lot 3); Anti-HPV 31; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; GMT ratio = 1.02, 95% CI 2-sided [0.90 to 1.15] — GMT ratio = GMT for 9- to 15-Year-Old Females (Lot 2) divided by GMT for 9- to 15-Year-Old Females (Lot 3)
Statistical Analysis 16: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Females (Lot 2); Anti-HPV 33; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; GMT ratio = 1.05, 95% CI 2-sided [0.94 to 1.16] — GMT ratio = GMT for 9- to 15-Year-Old Females (Lot 1) divided by GMT for 9- to 15-Year-Old Females (Lot 2)
Statistical Analysis 17: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Females (Lot 3); Anti-HPV 33; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; GMT ratio = 1.05, 95% CI 2-sided [0.94 to 1.17] — GMT ratio = GMT for 9- to 15-Year-Old Females (Lot 1) divided by GMT for 9- to 15-Year-Old Females (Lot 3)
Statistical Analysis 18: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 2) vs Base Study: 9- to 15-Year-Old Females (Lot 3); Anti-HPV 33; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; GMT ratio = 1.01, 95% CI 2-sided [0.90 to 1.12] — GMT ratio = GMT for 9- to 15-Year-Old Females (Lot 2) divided by GMT for 9- to 15-Year-Old Females (Lot 3)
Statistical Analysis 19: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Females (Lot 2); Anti-HPV 45; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; GMT ratio = 0.84, 95% CI 2-sided [0.73 to 0.95] — GMT ratio = GMT for 9- to 15-Year-Old Females (Lot 1) divided by GMT for 9- to 15-Year-Old Females (Lot 2)
Statistical Analysis 20: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Females (Lot 3); Anti-HPV 45; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; GMT ratio = 1.04, 95% CI 2-sided [0.91 to 1.18] — GMT ratio = GMT for 9- to 15-Year-Old Females (Lot 1) divided by GMT for 9- to 15-Year-Old Females (Lot 3)
Statistical Analysis 21: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 2) vs Base Study: 9- to 15-Year-Old Females (Lot 3); Anti-HPV 45; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; GMT ratio = 1.24, 95% CI 2-sided [1.08 to 1.42] — GMT ratio = GMT for 9- to 15-Year-Old Females (Lot 2) divided by GMT for 9- to 15-Year-Old Females (Lot 3)
Statistical Analysis 22: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Females (Lot 2); Anti-HPV 52; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; GMT ratio = 0.92, 95% CI 2-sided [0.83 to 1.03] — GMT ratio = GMT for 9- to 15-Year-Old Females (Lot 1) divided by GMT for 9- to 15-Year-Old Females (Lot 2)
Statistical Analysis 23: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Females (Lot 3); Anti-HPV 52; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; GMT ratio = 0.95, 95% CI 2-sided [0.85 to 1.07] — GMT ratio = GMT for 9- to 15-Year-Old Females (Lot 1) divided by GMT for 9- to 15-Year-Old Females (Lot 3)
Statistical Analysis 24: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 2) vs Base Study: 9- to 15-Year-Old Females (Lot 3); Anti-HPV 52; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; GMT ratio = 1.03, 95% CI 2-sided [0.92 to 1.16] — GMT ratio = GMT for 9- to 15-Year-Old Females (Lot 2) divided by GMT for 9- to 15-Year-Old Females (Lot 3)
Statistical Analysis 25: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Females (Lot 2); Anti-HPV 58; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; GMT ratio = 0.95, 95% CI 2-sided [0.86 to 1.06] — GMT ratio = GMT for 9- to 15-Year-Old Females (Lot 1) divided by GMT for 9- to 15-Year-Old Females (Lot 2)
Statistical Analysis 26: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Females (Lot 3); Anti-HPV 58; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; GMT ratio = 1.07, 95% CI 2-sided [0.96 to 1.20] — GMT ratio = GMT for 9- to 15-Year-Old Females (Lot 1) divided by GMT for 9- to 15-Year-Old Females (Lot 3)
Statistical Analysis 27: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 2) vs Base Study: 9- to 15-Year-Old Females (Lot 3); Anti-HPV 58; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; GMT ratio = 1.12, 95% CI 2-sided [1.00 to 1.26] — GMT ratio = GMT for 9- to 15-Year-Old Females (Lot 2) divided by GMT for 9- to 15-Year-Old Females (Lot 3)

4. Primary Outcome: Base Study: Percentage of Participants With Injection Site Adverse Experiences (AEs)
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study vaccine, whether or not considered related to the use of the vaccine. Any worsening of a preexisting condition which is temporally associated with the use of the study vaccine was also an AE. AEs such as redness, swelling, and pain/tenderness/soreness at the injection site were recorded.
Time Frame: Up to 5 days after any vaccination
Population: All participants who received at least one dose of 9vHPV vaccine and had available follow-up data. Per protocol, this outcome measure included data from 9- to 15-year-old females regardless of lot administered.
Measure: Number; unit: Percentage of Participants
Groups:
- 9- to 15-Year-Old Females (Lots 1, 2 or 3): 9-valent human papillomavirus (9vHPV) L1 VLP vaccine, 0.5 mL intramuscular injection at Day 1, Month 2, and Month 6. Vaccine dose administered is obtained from manufacturing Lots 1, 2, or 3.
Arm/Group | 9- to 15-Year-Old Females (Lots 1, 2 or 3) | Base Study: 9- to 15-Year-Old Males (Lot 1) | Base Study: 16- to 26-Year-Old Females (Lot 1)
Number analyzed (Participants) | 1923 | 662 | 466
Percentage of Participants | 81.9 | 72.8 | 85.4

5. Primary Outcome: Base Study: Percentage of Participants With Systemic AEs
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study vaccine, whether or not considered related to the use of the vaccine. Any worsening of a preexisting condition which is temporally associated with the use of the study vaccine was also an AE. Systemic AEs were those not categorized as injection-site AEs.
Time Frame: Up to 15 days after any vaccination
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | 9- to 15-Year-Old Females (Lots 1, 2 or 3) | Base Study: 9- to 15-Year-Old Males (Lot 1) | Base Study: 16- to 26-Year-Old Females (Lot 1)
Number analyzed (Participants) | 1923 | 662 | 466
Percentage of Participants | 45.0 | 41.8 | 57.1

6. Primary Outcome: Base Study: Percentage of Participants With Body Temperature ≥100.0°F (≥37.8ºC)
Description: Participants collected their oral body temperature in the evening of their vaccination day and at the same time each day thereafter for 4 days. The maximum body temperature obtained within 5 days of any of the 3 vaccinations was recorded. The percentage of participants who had at least 1 oral body temperature reading that was ≥100.0°F (≥37.8ºC) was summarized.
Time Frame: Up to 5 days after any vaccination
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Groups:
- 9- to 15-Year-Old Females (Lots 1, 2, or 3): Multivalent HPV L1 VLP vaccine, 0.5 mL intramuscular injection at Day 1, Month 2, and Month 6. Vaccine dose administered is obtained from manufacturing Lots 1, 2, or 3.
Arm/Group | 9- to 15-Year-Old Females (Lots 1, 2, or 3) | Base Study: 9- to 15-Year-Old Males (Lot 1) | Base Study: 16- to 26-Year-Old Females (Lot 1)
Number analyzed (Participants) | 1908 | 660 | 463
Percentage of Participants | 8.4 | 10.0 | 8.4

7. Secondary Outcome: Base Study: Percentage of Participants Who Seroconvert to Each of the HPV Types Contained in the Vaccine (9- to 15-Year-Old Females [Lot 1] and 16- to 26-Year-Old Females [Lot 1])
Description: Serum antibody titers for HPV virus-like particles (VLPs), Types 6, 11, 16, 18, 31, 33, 45, 52 and 58 were determined 4 weeks post-vaccination 3 using cLIA. The serostatus cutoffs (milli Merck U/mL) for HPV types were as follows: HPV Type 6: ≥30, HPV Type 11: ≥16; HPV Type 16: ≥20, HPV Type 18: ≥24, HPV Type 31: ≥10, HPV Type 33: ≥8, HPV Type 45: ≥8, HPV Type 52: ≥8, and HPV Type 58: ≥8.
Time Frame: 4 weeks post-vaccination 3 (Month 7)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Base Study: 9- to 15-Year-Old Females (Lot 1) | Base Study: 9- to 15-Year-Old Males (Lot 1)
Number analyzed (Participants) | 535 | 378
Percentage of Participants
  Anti-HPV 6 cLIA ≥30 mMU/mL: number analyzed (Participants) | 517 | 328
  Anti-HPV 6 cLIA ≥30 mMU/mL | 99.8 [98.9 to 100] | 99.7 [98.3 to 100]
  Anti-HPV 11 cLIA ≥16 mMU/mL: number analyzed (Participants) | 517 | 332
  Anti-HPV 11 cLIA ≥16 mMU/mL | 100 [99.3 to 100.0] | 100 [98.9 to 100.0]
  Anti-HPV 16 cLIA ≥20 mMU/mL: number analyzed (Participants) | 529 | 329
  Anti-HPV 16 cLIA ≥20 mMU/mL | 100 [99.3 to 100.0] | 100 [98.9 to 100.0]
  Anti-HPV 18 cLIA ≥24 mMU/mL: number analyzed (Participants) | 531 | 345
  Anti-HPV 18 cLIA ≥24 mMU/mL | 99.8 [99.0 to 100.0] | 99.7 [98.4 to 100.0]
  Anti-HPV 31 cLIA ≥10 mMU/mL: number analyzed (Participants) | 522 | 340
  Anti-HPV 31 cLIA ≥10 mMU/mL | 100.0 [99.3 to 100.0] | 99.7 [98.4 to 100.0]
  Anti-HPV 33 cLIA ≥8 mMU/mL: number analyzed (Participants) | 534 | 354
  Anti-HPV 33 cLIA ≥8 mMU/mL | 100.0 [99.3 to 100.0] | 99.7 [98.4 to 100.0]
  Anti-HPV 45 cLIA ≥8 mMU/mL: number analyzed (Participants) | 534 | 368
  Anti-HPV 45 cLIA ≥8 mMU/mL | 99.8 [99.0 to 100.0] | 99.5 [98.1 to 99.9]
  Anti-HPV 52 cLIA ≥8 mMU/mL: number analyzed (Participants) | 533 | 337
  Anti-HPV 52 cLIA ≥8 mMU/mL | 100.0 [99.3 to 100.0] | 99.7 [98.4 to 100.0]
  Anti-HPV 58 cLIA ≥8 mMU/mL: number analyzed (Participants) | 531 | 332
  Anti-HPV 58 cLIA ≥8 mMU/mL | 100.0 [99.3 to 100.0] | 100.0 [98.9 to 100.0]
Statistical Analysis 1: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Males (Lot 1); Anti-HPV 6; Test type: Non-Inferiority — Noninferiority is demonstrated if the lower limit of the 95% CI for the percentage point difference is greater than -5; p < 0.001, Miettinen and Nurminen; Percentage Point Difference = 0.1, 95% CI 2-sided [-0.8 to 1.5] — Percentage Point Difference = 9- to 15-Year-Old Females (Lot 1) minus 16- to 26-Year-Old Females (Lot 1)
Statistical Analysis 2: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Males (Lot 1); Anti-HPV 11; Test type: Non-Inferiority — Noninferiority is demonstrated if the lower limit of the 95% CI for the percentage point difference is greater than -5; p < 0.001, Miettinen and Nurminen; Percentage Point Difference = 0.0, 95% CI 2-sided [-0.7 to 1.2] — Percentage Point Difference = 9- to 15-Year-Old Females (Lot 1) minus 16- to 26-Year-Old Females (Lot 1)
Statistical Analysis 3: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Males (Lot 1); Anti-HPV 16; Test type: Non-Inferiority — Noninferiority is demonstrated if the lower limit of the 95% CI for the percentage point difference is greater than -5; p < 0.001, Miettinen and Nurminen; Percentage Point Difference = 0.0, 95% CI 2-sided [-0.7 to 1.2] — Percentage Point Difference = 9- to 15-Year-Old Females (Lot 1) minus 16- to 26-Year-Old Females (Lot 1)
Statistical Analysis 4: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Males (Lot 1); Anti-HPV 18; Test type: Non-Inferiority — Noninferiority is demonstrated if the lower limit of the 95% CI for the percentage point difference is greater than -5; p < 0.001, Miettinen and Nurminen; Percentage Point Difference = 0.1, 95% CI 2-sided [-0.8 to 1.5] — Percentage Point Difference = 9- to 15-Year-Old Females (Lot 1) minus 16- to 26-Year-Old Females (Lot 1)
Statistical Analysis 5: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Males (Lot 1); Anti-HPV 31; Test type: Non-Inferiority — Noninferiority is demonstrated if the lower limit of the 95% CI for the percentage point difference is greater than -5; p < 0.001, Miettinen and Nurminen; Percentage Point Difference = 0.3, 95% CI 2-sided [-0.4 to 1.7] — Percentage Point Difference = 9- to 15-Year-Old Females (Lot 1) minus 16- to 26-Year-Old Females (Lot 1)
Statistical Analysis 6: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Males (Lot 1); Anti-HPV 33; Test type: Non-Inferiority — Noninferiority is demonstrated if the lower limit of the 95% CI for the percentage point difference is greater than -5; p < 0.001, Miettinen and Nurminen; Percentage Point Difference = 0.3, 95% CI 2-sided [-0.4 to 1.6] — Percentage Point Difference = 9- to 15-Year-Old Females (Lot 1) minus 16- to 26-Year-Old Females (Lot 1)
Statistical Analysis 7: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Males (Lot 1); Anti-HPV 45; Test type: Non-Inferiority — Noninferiority is demonstrated if the lower limit of the 95% CI for the percentage point difference is greater than -5; p < 0.001, Miettinen and Nurminen; Percentage Point Difference = 0.4, 95% CI 2-sided [-0.6 to 1.8] — Percentage Point Difference = 9- to 15-Year-Old Females (Lot 1) minus 16- to 26-Year-Old Females (Lot 1)
Statistical Analysis 8: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Males (Lot 1); Anti-HPV 52; Test type: Non-Inferiority — Noninferiority is demonstrated if the lower limit of the 95% CI for the percentage point difference is greater than -5; p < 0.001, Miettinen and Nurminen; Percentage Point Difference = 0.3, 95% CI 2-sided [-0.4 to 1.7] — Percentage Point Difference = 9- to 15-Year-Old Females (Lot 1) minus 16- to 26-Year-Old Females (Lot 1)
Statistical Analysis 9: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Males (Lot 1); Anti-HPV 58; Test type: Non-Inferiority — Noninferiority is demonstrated if the lower limit of the 95% CI for the percentage point difference is greater than -5; p < 0.001, Miettinen and Nurminen; Percentage Point Difference = 0.0, 95% CI 2-sided [-0.7 to 1.2] — Percentage Point Difference = 9- to 15-Year-Old Females (Lot 1) minus 16- to 26-Year-Old Females (Lot 1)

8. Secondary Outcome: Base Study: Percentage of Participants Who Seroconvert to Each of the HPV Types Contained in the Vaccine (9- to 15-Year-Old Males [Lot 1] Versus 16- to 26-Year-Old Females [Lot 1])
Description: Serum antibody titers for HPV VLPs, Types 6, 11, 16, 18, 31, 33, 45, 52 and 58 were determined 4 weeks post-vaccination 3 using cLIA. The serostatus cutoffs (milli Merck U/mL) for HPV types were as follows: HPV Type 6: ≥30, HPV Type 11: ≥16; HPV Type 16: ≥20, HPV Type 18: ≥24, HPV Type 31: ≥10, HPV Type 33: ≥8, HPV Type 45: ≥8, HPV Type 52: ≥8, and HPV Type 58: ≥8.
Time Frame: 4 weeks post-vaccination 3 (Month 7)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Base Study: 9- to 15-Year-Old Males (Lot 1) | Base Study: 16- to 26-Year-Old Females (Lot 1)
Number analyzed (Participants) | 570 | 378
Percentage of Participants
  Anti-HPV 6 cLIA ≥30 mMU/mL: number analyzed (Participants) | 559 | 328
  Anti-HPV 6 cLIA ≥30 mMU/mL | 99.8 [99.0 to 100.0] | 99.7 [98.3 to 100.0]
  Anti-HPV 11 cLIA ≥16 mMU/mL: number analyzed (Participants) | 559 | 332
  Anti-HPV 11 cLIA ≥16 mMU/mL | 100.0 [99.3 to 100.0] | 100.0 [98.9 to 100.0]
  Anti-HPV 16 cLIA ≥20 mMU/mL: number analyzed (Participants) | 569 | 329
  Anti-HPV 16 cLIA ≥20 mMU/mL | 100.0 [99.4 to 100.0] | 100.0 [98.9 to 100.0]
  Anti-HPV 18 cLIA ≥24 mMU/mL: number analyzed (Participants) | 567 | 345
  Anti-HPV 18 cLIA ≥24 mMU/mL | 100.0 [99.4 to 100.0] | 99.7 [98.4 to 100.0]
  Anti-HPV 31 cLIA ≥10 mMU/mL: number analyzed (Participants) | 564 | 340
  Anti-HPV 31 cLIA ≥10 mMU/mL | 100.0 [99.3 to 100.0] | 99.7 [98.4 to 100.0]
  Anti-HPV 33 cLIA ≥8 mMU/mL: number analyzed (Participants) | 567 | 354
  Anti-HPV 33 cLIA ≥8 mMU/mL | 100.0 [99.4 to 100.0] | 99.7 [98.4 to 100.0]
  Anti-HPV 45 cLIA ≥8 mMU/mL: number analyzed (Participants) | 570 | 368
  Anti-HPV 45 cLIA ≥8 mMU/mL | 100.0 [99.4 to 100.0] | 99.5 [98.1 to 99.9]
  Anti-HPV 52 cLIA ≥8 mMU/mL: number analyzed (Participants) | 568 | 337
  Anti-HPV 52 cLIA ≥8 mMU/mL | 100.0 [99.4 to 100.0] | 99.7 [98.4 to 100.0]
  Anti-HPV 58 cLIA ≥8 mMU/mL: number analyzed (Participants) | 566 | 332
  Anti-HPV 58 cLIA ≥8 mMU/mL | 100.0 [99.4 to 100.0] | 100.0 [98.9 to 100.0]
Statistical Analysis 1: Comparison: Base Study: 9- to 15-Year-Old Males (Lot 1) vs Base Study: 16- to 26-Year-Old Females (Lot 1); Anti-HPV 6; Test type: Non-Inferiority — Noninferiority is demonstrated if the lower limit of the 95% CI for the percentage point difference is greater than -5; p < 0.001, Miettinen and Nurminen; Percentage Point Difference = 0.1, 95% CI 2-sided [-0.7 to 1.5] — Percentage Point Difference = 9- to 15-Year-Old Males (Lot 1) minus 16- to 26-Year-Old Females (Lot 1)
Statistical Analysis 2: Comparison: Base Study: 9- to 15-Year-Old Males (Lot 1) vs Base Study: 16- to 26-Year-Old Females (Lot 1); Anti-HPV 11; Test type: Non-Inferiority — Noninferiority is demonstrated if the lower limit of the 95% CI for the percentage point difference is greater than -5; p < 0.001, Miettinen and Nurminen; Percentage Point Difference = 0.0, 95% CI 2-sided [-0.7 to 1.2] — Percentage Point Difference = 9- to 15-Year-Old Males (Lot 1) minus 16- to 26-Year-Old Females (Lot 1)
Statistical Analysis 3: Comparison: Base Study: 9- to 15-Year-Old Males (Lot 1) vs Base Study: 16- to 26-Year-Old Females (Lot 1); Anti-HPV 16; Test type: Non-Inferiority — Noninferiority is demonstrated if the lower limit of the 95% CI for the percentage point difference is greater than -5; p < 0.001, Miettinen and Nurminen; Percentage Point Difference = 0.0, 95% CI 2-sided [-0.7 to 1.2] — Percentage Point Difference = 9- to 15-Year-Old Males (Lot 1) minus 16- to 26-Year-Old Females (Lot 1)
Statistical Analysis 4: Comparison: Base Study: 9- to 15-Year-Old Males (Lot 1) vs Base Study: 16- to 26-Year-Old Females (Lot 1); Anti-HPV 18; Test type: Non-Inferiority — Noninferiority is demonstrated if the lower limit of the 95% CI for the percentage point difference is greater than -5; p < 0.001, Miettinen and Nurminen; Percentage Point Difference = 0.3, 95% CI 2-sided [-0.4 to 1.6] — Percentage Point Difference = 9- to 15-Year-Old Males (Lot 1) minus 16- to 26-Year-Old Females (Lot 1)
Statistical Analysis 5: Comparison: Base Study: 9- to 15-Year-Old Males (Lot 1) vs Base Study: 16- to 26-Year-Old Females (Lot 1); Anti-HPV 31; Test type: Non-Inferiority — Noninferiority is demonstrated if the lower limit of the 95% CI for the percentage point difference is greater than -5; p < 0.001, Miettinen and Nurminen; Percentage Point Difference = 0.3, 95% CI 2-sided [-0.4 to 1.7] — Percentage Point Difference = 9- to 15-Year-Old Males (Lot 1) minus 16- to 26-Year-Old Females (Lot 1)
Statistical Analysis 6: Comparison: Base Study: 9- to 15-Year-Old Males (Lot 1) vs Base Study: 16- to 26-Year-Old Females (Lot 1); Anti-HPV 33; Test type: Non-Inferiority — Noninferiority is demonstrated if the lower limit of the 95% CI for the percentage point difference is greater than -5; p < 0.001, Miettinen and Nurminen; Percentage Point Difference = 0.3, 95% CI 2-sided [-0.4 to 1.6] — Percentage Point Difference = 9- to 15-Year-Old Males (Lot 1) minus 16- to 26-Year-Old Females (Lot 1)
Statistical Analysis 7: Comparison: Base Study: 9- to 15-Year-Old Males (Lot 1) vs Base Study: 16- to 26-Year-Old Females (Lot 1); Anti-HPV 45; Test type: Non-Inferiority — Noninferiority is demonstrated if the lower limit of the 95% CI for the percentage point difference is greater than -5; p < 0.001, Miettinen and Nurminen; Percentage Point Difference = 0.5, 95% CI 2-sided [-0.1 to 2.0] — Percentage Point Difference = 9- to 15-Year-Old Males (Lot 1) minus 16- to 26-Year-Old Females (Lot 1)
Statistical Analysis 8: Comparison: Base Study: 9- to 15-Year-Old Males (Lot 1) vs Base Study: 16- to 26-Year-Old Females (Lot 1); Anti-HPV 52; Test type: Non-Inferiority — Noninferiority is demonstrated if the lower limit of the 95% CI for the percentage point difference is greater than -5; p < 0.001, Miettinen and Nurminen; Percentage Point Difference = 0.3, 95% CI 2-sided [-0.4 to 1.7] — Percentage Point Difference = 9- to 15-Year-Old Males (Lot 1) minus 16- to 26-Year-Old Females (Lot 1)
Statistical Analysis 9: Comparison: Base Study: 9- to 15-Year-Old Males (Lot 1) vs Base Study: 16- to 26-Year-Old Females (Lot 1); Anti-HPV 58; Test type: Non-Inferiority — Noninferiority is demonstrated if the lower limit of the 95% CI for the percentage point difference is greater than -5; p < 0.001, Miettinen and Nurminen; Percentage Point Difference = 0.0, 95% CI 2-sided [-0.7 to 1.2] — Percentage Point Difference = 9- to 15-Year-Old Males (Lot 1) minus 16- to 26-Year-Old Females (Lot 1)

9. Secondary Outcome: Base Study: Percentage of Participants Who Seroconvert to Each of the HPV Types Contained in the Vaccine (Lot Consistency Study)
Description: Serum antibody titers for HPV virus-like particles (VLPs), Types 6, 11, 16, 18, 31, 33, 45, 52 and 58 were determined 4 weeks post- vaccination 3 using cLIA. The serostatus cutoffs (milli Merck U/mL) for HPV types were as follows: HPV Type 6: ≥30, HPV Type 11: ≥16; HPV Type 16: ≥20, HPV Type 18: ≥24, HPV Type 31: ≥10, HPV Type 33: ≥8, HPV Type 45: ≥8, HPV Type 52: ≥8, and HPV Type 58: ≥8.
Time Frame: 4 weeks post-vaccination 3 (Month 7)
Population: 9- to 15-year-old females who received 3 vaccinations from Lots 1, 2, and 3 and met following criteria for at least 1 of the 9 HPV types: no general protocol violations, received all 3 vaccinations within acceptable day ranges, seronegative at Day 1 for HPV type(s), and had a Month 7 serum sample collected within an acceptable day range
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Base Study: 9- to 15-Year-Old Females (Lot 1) | Base Study: 9- to 15-Year-Old Females (Lot 2) | Base Study: 9- to 15-Year-Old Females (Lot 3)
Number analyzed (Participants) | 535 | 549 | 565
Percentage of Participants
  HPV 6 cLIA ≥30 mMU/mL: number analyzed (Participants) | 517 | 536 | 544
  HPV 6 cLIA ≥30 mMU/mL | 99.8 [98.9 to 100.0] | 99.8 [99.0 to 100.0] | 99.3 [98.1 to 99.8]
  HPV 11 cLIA ≥16 mMU/mL: number analyzed (Participants) | 517 | 536 | 544
  HPV 11 cLIA ≥16 mMU/mL | 100.0 [99.3 to 100.0] | 100.0 [99.3 to 100.0] | 99.6 [98.7 to 100.0]
  HPV 16 cLIA ≥20 mMU/mL: number analyzed (Participants) | 529 | 542 | 556
  HPV 16 cLIA ≥20 mMU/mL | 100.0 [99.3 to 100.0] | 100.0 [99.3 to 100.0] | 99.6 [98.7 to 100.0]
  HPV 18 cLIA ≥24 mMU/mL: number analyzed (Participants) | 531 | 547 | 563
  HPV 18 cLIA ≥24 mMU/mL | 99.8 [99.0 to 100.0] | 100.0 [99.3 to 100.0] | 99.6 [98.7 to 100.0]
  HPV 31 cLIA ≥10 mMU/mL: number analyzed (Participants) | 522 | 542 | 553
  HPV 31 cLIA ≥10 mMU/mL | 100.0 [99.3 to 100.0] | 100.0 [99.3 to 100.0] | 99.8 [99.0 to 100.0]
  HPV 33 cLIA ≥8 mMU/mL: number analyzed (Participants) | 534 | 543 | 560
  HPV 33 cLIA ≥8 mMU/mL | 100.0 [99.3 to 100.0] | 100.0 [99.3 to 100.0] | 99.6 [98.7 to 100.0]
  HPV 45 cLIA ≥8 mMU/mL: number analyzed (Participants) | 534 | 548 | 565
  HPV 45 cLIA ≥8 mMU/mL | 99.8 [99.0 to 100.0] | 100.0 [99.3 to 100.0] | 99.6 [98.7 to 100.0]
  HPV 52 cLIA ≥8 mMU/mL: number analyzed (Participants) | 533 | 547 | 562
  HPV 52 cLIA ≥8 mMU/mL | 100.0 [99.3 to 100.0] | 100.0 [99.3 to 100.0] | 99.6 [98.7 to 100.0]
  HPV 58 cLIA ≥8 mMU/mL: number analyzed (Participants) | 531 | 539 | 560
  HPV 58 cLIA ≥8 mMU/mL | 100.0 [99.3 to 100.0] | 100.0 [99.3 to 100.0] | 99.6 [98.7 to 100.0]
Statistical Analysis 1: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Females (Lot 2); Anti-HPV 6; Test type: Equivalence — equivalence requires that the two-sided 95% CI for the difference in percentages between lots be entirely contained within the interval (-5, 5); Percentage Point Difference = 0.0, 95% CI 2-sided [-0.9 to 0.9] — Percentage Point Difference = 9- to 15-Year-Old Females (Lot 1) minus 9- to 15-Year-Old Females (Lot 2)
Statistical Analysis 2: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Females (Lot 3); Anti-HPV 6; Test type: Equivalence — [test comment as in outcome 9, analysis 1]; Percentage Point Difference = 0.5, 95% CI 2-sided [-0.4 to 1.7] — Percentage Point Difference = 9- to 15-Year-Old Females (Lot 1) minus 9- to 15-Year-Old Females (Lot 3)
Statistical Analysis 3: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 2) vs Base Study: 9- to 15-Year-Old Females (Lot 3); Anti-HPV 6; Test type: Equivalence — [test comment as in outcome 9, analysis 1]; Percentage Point Difference = 0.6, 95% CI 2-sided [-0.4 to 1.7] — Percentage Point Difference = 9- to 15-Year-Old Females (Lot 2) minus 9- to 15-Year-Old Females (Lot 3)
Statistical Analysis 4: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Females (Lot 2); Anti-HPV 11; Test type: Equivalence — [test comment as in outcome 9, analysis 1]; Percentage Point Difference = 0.0, 95% CI 2-sided [-0.7 to 0.7] — Percentage Point Difference = 9- to 15-Year-Old Females (Lot 1) minus 9- to 15-Year-Old Females (Lot 2)
Statistical Analysis 5: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Females (Lot 3); Anti-HPV 11; Test type: Equivalence — [test comment as in outcome 9, analysis 1]; Percentage Point Difference = 0.4, 95% CI 2-sided [-0.4 to 1.3] — Percentage Point Difference = 9- to 15-Year-Old Females (Lot 1) minus 9- to 15-Year-Old Females (Lot 3)
Statistical Analysis 6: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 2) vs Base Study: 9- to 15-Year-Old Females (Lot 3); Anti-HPV 11; Test type: Equivalence — [test comment as in outcome 9, analysis 1]; Percentage Point Difference = 0.4, 95% CI 2-sided [-0.4 to 1.3] — Percentage Point Difference = 9- to 15-Year-Old Females (Lot 2) minus 9- to 15-Year-Old Females (Lot 3)
Statistical Analysis 7: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Females (Lot 2); Anti-HPV 16; Test type: Equivalence — [test comment as in outcome 9, analysis 1]; Percentage Point Difference = 0.0, 95% CI 2-sided [-0.7 to 0.7] — Percentage Point Difference = 9- to 15-Year-Old Females (Lot 1) minus 9- to 15-Year-Old Females (Lot 2)
Statistical Analysis 8: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Females (Lot 3); Anti-HPV 16; Test type: Equivalence — [test comment as in outcome 9, analysis 1]; Percentage Point Difference = 0.4, 95% CI 2-sided [-0.4 to 1.3] — Percentage Point Difference = 9- to 15-Year-Old Females (Lot 1) minus 9- to 15-Year-Old Females (Lot 3)
Statistical Analysis 9: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 2) vs Base Study: 9- to 15-Year-Old Females (Lot 3); Anti-HPV 16; Test type: Equivalence — [test comment as in outcome 9, analysis 1]; Percentage Point Difference = 0.4, 95% CI 2-sided [-0.4 to 1.3] — Percentage Point Difference = 9- to 15-Year-Old Females (Lot 2) minus 9- to 15-Year-Old Females (Lot 3)
Statistical Analysis 10: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Females (Lot 2); Anti-HPV 18; Test type: Equivalence — [test comment as in outcome 9, analysis 1]; Percentage Point Difference = -0.2, 95% CI 2-sided [-1.1 to 0.5] — Percentage Point Difference = 9- to 15-Year-Old Females (Lot 1) minus 9- to 15-Year-Old Females (Lot 2)
Statistical Analysis 11: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Females (Lot 3); Anti-HPV 18; Test type: Equivalence — [test comment as in outcome 9, analysis 1]; Percentage Point Difference = 0.2, 95% CI 2-sided [-0.7 to 1.1] — Percentage Point Difference = 9- to 15-Year-Old Females (Lot 1) minus 9- to 15-Year-Old Females (Lot 3)
Statistical Analysis 12: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 2) vs Base Study: 9- to 15-Year-Old Females (Lot 3); Anti-HPV 18; Test type: Equivalence — [test comment as in outcome 9, analysis 1]; Percentage Point Difference = 0.4, 95% CI 2-sided [-0.4 to 1.3] — Percentage Point Difference = 9- to 15-Year-Old Females (Lot 2) minus 9- to 15-Year-Old Females (Lot 3)
Statistical Analysis 13: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Females (Lot 2); Anti-HPV 31; Test type: Equivalence — [test comment as in outcome 9, analysis 1]; Percentage Point Difference = 0.0, 95% CI 2-sided [-0.7 to 0.7] — Percentage Point Difference = 9- to 15-Year-Old Females (Lot 1) minus 9- to 15-Year-Old Females (Lot 2)
Statistical Analysis 14: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Females (Lot 3); Anti-HPV 31; Test type: Equivalence — [test comment as in outcome 9, analysis 1]; Percentage Point Difference = 0.2, 95% CI 2-sided [-0.6 to 1.0] — Percentage Point Difference = 9- to 15-Year-Old Females (Lot 1) minus 9- to 15-Year-Old Females (Lot 3)
Statistical Analysis 15: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 2) vs Base Study: 9- to 15-Year-Old Females (Lot 3); Anti-HPV 31; Test type: Equivalence — [test comment as in outcome 9, analysis 1]; Percentage Point Difference = 0.2, 95% CI 2-sided [-0.5 to 1.0] — Percentage Point Difference = 9- to 15-Year-Old Females (Lot 2) minus 9- to 15-Year-Old Females (Lot 3)
Statistical Analysis 16: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Females (Lot 2); Anti-HPV 33; Test type: Equivalence — [test comment as in outcome 9, analysis 1]; Percentage Point Difference = 0.0, 95% CI 2-sided [-0.7 to 0.7] — Percentage Point Difference = 9- to 15-Year-Old Females (Lot 1) minus 9- to 15-Year-Old Females (Lot 2)
Statistical Analysis 17: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Females (Lot 3); Anti-HPV 33; Test type: Equivalence — [test comment as in outcome 9, analysis 1]; Percentage Point Difference = 0.4, 95% CI 2-sided [-0.4 to 1.3] — Percentage Point Difference = 9- to 15-Year-Old Females (Lot 1) minus 9- to 15-Year-Old Females (Lot 3)
Statistical Analysis 18: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 2) vs Base Study: 9- to 15-Year-Old Females (Lot 3); Anti-HPV 33; Test type: Equivalence — [test comment as in outcome 9, analysis 1]; Percentage Point Difference = 0.4, 95% CI 2-sided [-0.4 to 1.3] — Percentage Point Difference = 9- to 15-Year-Old Females (Lot 2) minus 9- to 15-Year-Old Females (Lot 3)
Statistical Analysis 19: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Females (Lot 2); Anti-HPV 45; Test type: Equivalence — [test comment as in outcome 9, analysis 1]; Percentage Point Difference = -0.2, 95% CI 2-sided [-1.1 to 0.5] — Percentage Point Difference = 9- to 15-Year-Old Females (Lot 1) minus 9- to 15-Year-Old Females (Lot 2)
Statistical Analysis 20: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Females (Lot 3); Anti-HPV 45; Test type: Equivalence — [test comment as in outcome 9, analysis 1]; Percentage Point Difference = 0.2, 95% CI 2-sided [-0.7 to 1.1] — Percentage Point Difference = 9- to 15-Year-Old Females (Lot 1) minus 9- to 15-Year-Old Females (Lot 3)
Statistical Analysis 21: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 2) vs Base Study: 9- to 15-Year-Old Females (Lot 3); Anti-HPV 45; Test type: Equivalence — [test comment as in outcome 9, analysis 1]; Percentage Point Difference = 0.4, 95% CI 2-sided [-0.4 to 1.3] — Percentage Point Difference = 9- to 15-Year-Old Females (Lot 2) minus 9- to 15-Year-Old Females (Lot 3)
Statistical Analysis 22: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Females (Lot 2); Anti-HPV 52; Test type: Equivalence — [test comment as in outcome 9, analysis 1]; Percentage Point Difference = 0.0, 95% CI 2-sided [-0.7 to 0.7] — Percentage Point Difference = 9- to 15-Year-Old Females (Lot 1) minus 9- to 15-Year-Old Females (Lot 2)
Statistical Analysis 23: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Females (Lot 3); Anti-HPV 52; Test type: Equivalence — [test comment as in outcome 9, analysis 1]; Percentage Point Difference = 0.3, 95% CI 2-sided [-0.4 to 1.3] — Percentage Point Difference = 9- to 15-Year-Old Females (Lot 1) minus 9- to 15-Year-Old Females (Lot 3)
Statistical Analysis 24: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 2) vs Base Study: 9- to 15-Year-Old Females (Lot 3); Anti-HPV 52; Test type: Equivalence — [test comment as in outcome 9, analysis 1]; Percentage Point Difference = 0.4, 95% CI 2-sided [-0.4 to 1.3] — Percentage Point Difference = 9- to 15-Year-Old Females (Lot 2) minus 9- to 15-Year-Old Females (Lot 3)
Statistical Analysis 25: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Females (Lot 2); Anti-HPV 58; Test type: Equivalence — [test comment as in outcome 9, analysis 1]; Percentage Point Difference = 0.0, 95% CI 2-sided [-0.7 to 0.7] — Percentage Point Difference = 9- to 15-Year-Old Females (Lot 1) minus 9- to 15-Year-Old Females (Lot 2)
Statistical Analysis 26: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 1) vs Base Study: 9- to 15-Year-Old Females (Lot 3); Anti-HPV 58; Test type: Equivalence — [test comment as in outcome 9, analysis 1]; Percentage Point Difference = 0.4, 95% CI 2-sided [-0.4 to 1.3] — Percentage Point Difference = 9- to 15-Year-Old Females (Lot 1) minus 9- to 15-Year-Old Females (Lot 3)
Statistical Analysis 27: Comparison: Base Study: 9- to 15-Year-Old Females (Lot 2) vs Base Study: 9- to 15-Year-Old Females (Lot 3); Anti-HPV 58; Test type: Equivalence — [test comment as in outcome 9, analysis 1]; Percentage Point Difference = 0.4, 95% CI 2-sided [-0.4 to 1.3] — Percentage Point Difference = 9- to 15-Year-Old Females (Lot 2) minus 9- to 15-Year-Old Females (Lot 3)

10. Primary Outcome: Extension Study: GMTs For Each of the HPV Types Contained in the Vaccine
Description: Serum antibody titers (milli Merck Units/mL) measured by cLIA to each of the 9vHPV types were assessed. Per protocol, the extension study included data from 9- to 15-year-old females regardless of lot administered.
Time Frame: Up to ~Month 126
Population: All participants who met the following criteria for at least 1 of the 9 HPV types: no general protocol violations, received all 3 vaccinations within acceptable day ranges, seronegative at Day 1 for HPV type(s), and had a Month 7 serum sample collected within an acceptable day range.
Measure: Geometric Mean (95% Confidence Interval); unit: milli Merck Units/mL
Arm/Group | Extension Study: 9- to 15-Year-Old Females | Extension Study: 9- to 15-Year-Old Males
Number analyzed (Participants) | 971 | 301
milli Merck Units/mL
  Anti-HPV 6: number analyzed (Participants) | 341 | 176
  Anti-HPV 6 | 122.3 [111.1 to 134.7] | 129.5 [112.5 to 149.1]
  Anti-HPV 11: number analyzed (Participants) | 332 | 169
  Anti-HPV 11 | 80.2 [72.5 to 88.8] | 91.0 [78.4 to 105.6]
  Anti-HPV 16: number analyzed (Participants) | 388 | 173
  Anti-HPV 16 | 403.0 [357.3 to 454.5] | 414.3 [353.8 to 485.3]
  Anti-HPV 18: number analyzed (Participants) | 347 | 178
  Anti-HPV 18 | 128.1 [116.7 to 140.7] | 148.4 [130.2 to 169.2]
  Anti-HPV 31: number analyzed (Participants) | 343 | 177
  Anti-HPV 31 | 108.9 [97.6 to 121.6] | 128.6 [111.2 to 148.8]
  Anti-HPV 33: number analyzed (Participants) | 344 | 178
  Anti-HPV 33 | 59.2 [53.7 to 65.2] | 69.6 [60.7 to 79.7]
  Anti-HPV 45: number analyzed (Participants) | 325 | 169
  Anti-HPV 45 | 42.1 [37.7 to 47.1] | 49.8 [43.0 to 57.8]
  Anti-HPV 52: number analyzed (Participants) | 348 | 176
  Anti-HPV 52 | 55.3 [50.5 to 60.6] | 59.6 [52.0 to 68.4]
  Anti-HPV 58: number analyzed (Participants) | 342 | 175
  Anti-HPV 58 | 76.5 [69.2 to 84.6] | 90.5 [78.4 to 104.6]

11. Primary Outcome: Extension Study: Percentage of Participants Who Are Seropositive to Each of the HPV Types Contained in the Vaccine
Description: Serum antibody titers for HPV VLPs Types 6, 11, 16, 18, 31, 33, 45, 52 and 58 was determined and reported in milli Merck Units/mL. The percentage of participants seropositive to each HPV type was reported. Per protocol, the extension study included data from 9- to 15-year-old females regardless of lot administered.
Time Frame: Up to ~Month 126
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Extension Study: 9- to 15-Year-Old Females | Extension Study: 9- to 15-Year-Old Males
Number analyzed (Participants) | 971 | 301
Percentage of Participants
  Anti-HPV 6: number analyzed (Participants) | 341 | 176
  Anti-HPV 6 | 82.7 [78.3 to 86.6] | 84.1 [77.8 to 89.2]
  Anti-HPV 11: number analyzed (Participants) | 332 | 169
  Anti-HPV 11 | 85.2 [81.0 to 88.9] | 87.0 [81.0 to 91.7]
  Anti-HPV 16: number analyzed (Participants) | 338 | 173
  Anti-HPV 16 | 97.3 [95.0 to 98.8] | 98.3 [95.0 to 99.6]
  Anti-HPV 18: number analyzed (Participants) | 347 | 178
  Anti-HPV 18 | 80.1 [75.5 to 84.2] | 83.7 [77.4 to 88.8]
  Anti-HPV 31: number analyzed (Participants) | 343 | 177
  Anti-HPV 31 | 90.1 [86.4 to 93.0] | 92.7 [87.8 to 96.0]
  Anti-HPV 33: number analyzed (Participants) | 344 | 178
  Anti-HPV 33 | 85.2 [81.0 to 88.8] | 89.3 [83.8 to 93.4]
  Anti-HPV 45: number analyzed (Participants) | 325 | 169
  Anti-HPV 45 | 81.8 [77.2 to 85.9] | 92.3 [87.2 to 95.8]
  Anti-HPV 52: number analyzed (Participants) | 348 | 176
  Anti-HPV 52 | 88.2 [84.4 to 91.4] | 89.2 [83.7 to 93.4]
  Anti-HPV 58: number analyzed (Participants) | 342 | 175
  Anti-HPV 58 | 96.5 [94.0 to 98.2] | 97.1 [93.5 to 99.1]

12. Secondary Outcome: Extension Study: Combined Incidence of HPV 6/11/16/18/31/33/45/52/58-Related Persistent Infection in Females
Description: Persistent infection is when a participant is positive by polymerase chain reaction (PCR) for the same HPV type in cervicovaginal/external genital swabs or tissue specimens collected at consecutive visits at least 6 months (+/-1 month visit window) apart. Incidence was estimated as cases per 10,000 person-years. Person-years follow-up was from beginning of long-term follow-up or when a study participant reached 16 years of age, whichever came later. Per protocol, the extension study included 9- to 15-year-old females regardless of lot administered.
Time Frame: Up to ~Month 126
Population: The per-protocol effectiveness population, which included participants who were seronegative (by cLIA) to the relevant HPV type(s) at Day 1 (seronegative to both HPV 6 and 11 for analysis of HPV 6 and 11 HPV11-related endpoints), received all 3 doses of 9vHPV vaccine with the correct dose of the clinical material within 1 year, and had no other protocol violation that could interfere with evaluation of vaccine effectiveness.
Measure: Number (95% Confidence Interval); unit: Cases per 10,000 person-years
Arm/Group | Extension Study: 9- to 15-Year-Old Females
Number analyzed (Participants) | 872
Cases per 10,000 person-years | 52.4 (33.6) [33.6 to 78.0]

13. Secondary Outcome: Extension Study: Combined Incidence of HPV 6/11/16/18/31/33/45/52/58-Related Persistent Infection in Males
Description: Persistent infection is when a participant is positive by PCR for the same HPV type in external genital swabs or tissue specimens collected at consecutive visits at least 6 months (+/-1 month visit window) apart. Incidence was estimated as cases per 10,000 person-years. Person-years follow-up was from beginning of long-term follow-up or when a study participant reached 16 years of age, whichever came later.
Time Frame: Up to ~Month 126
Population: The per-protocol effectiveness population, which included participants who were seronegative (by cLIA) to the relevant HPV type(s) at Day 1 (seronegative to both HPV 6 and 11 for analysis of HPV 6 and 11-related endpoints), received all 3 doses of 9vHPV vaccine with the correct dose of the clinical material within 1 year, and had no other protocol violation that could interfere with evaluation of vaccine effectiveness.
Measure: Number (95% Confidence Interval); unit: Cases per 10,000 person-years
Arm/Group | Extension Study: 9- to 15-Year-Old Males
Number analyzed (Participants) | 261
Cases per 10,000 person-years | 54.6 (21.9) [21.9 to 112.4]

14. Secondary Outcome: Extension Study: Combined Incidence of Cervical Intraepithelial Neoplasia, Vulvar Intraepithelial Neoplasia, Vaginal Intraepithelial Neoplasia, Genital Warts, and Cervical/Vulvar/Vaginal Cancers Related to HPV 6/11/16/18/31/33/45/52/58 in Females
Description: The combined incidence of cervical intraepithelial neoplasia, vulvar intraepithelial neoplasia, vaginal intraepithelial neoplasia, genital warts, and cervical/vulvar/vaginal cancers, related to HPV 6/11/16/18/31/33/45/52/58 was assessed. This outcome measure was determined by clinical/pathologic criteria and positive PCR assay for HPV type. Incidence was estimated as cases per 10,000 person-years. Person-years follow-up was calculated starting from the beginning of the long-term follow-up study or the date when the study participant reached 16 years of age, whichever came later. Per protocol, the extension study included data from 9- to 15-year-old females regardless of lot administered.
Time Frame: Up to ~Month 126
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: Cases per 10,000 person-years
Arm/Group | Extension Study: 9- to 15-Year-Old Females
Number analyzed (Participants) | 866
Cases per 10,000 person-years | 2.2 (0.1) [0.1 to 12.2]

15. Secondary Outcome: Extension Study: Combined Incidence of Penile Intraepithelial Neoplasia, Penile/Perineal/Perianal Cancers and Genital Warts Related to HPV 6/11/16/18/31/33/45/52/58 in Males
Description: The combined incidence of penile intraepithelial neoplasia, penile/perineal/perianal cancers, and genital warts related to HPV6/11/16/18/31/33/45/52/58 was assessed. This outcome measure was determined by clinical/pathologic criteria and positive PCR assay for HPV type. Incidence was estimated as cases per 10,000 person-years. For each study participant, person-years follow up was calculated starting from the beginning of the long-term follow-up study or the date when the study participant reached 16 years of age, whichever came later.
Time Frame: Up to ~Month 126
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: Cases per 10,000 person-years
Arm/Group | Extension Study: 9- to 15-Year-Old Males
Number analyzed (Participants) | 261
Cases per 10,000 person-years | 0.0 (0.0) [0.0 to 28.9]

16. Secondary Outcome: Extension Study: Percentage of Participants With Vaccine-Related or Procedure-Related Serious Adverse Events
Description: A serious adverse event (SAE) included a death which resulted in the participant discontinuing the study, a serious adverse experience that was considered by an investigator who was a qualified physician to be possibly, probably, or definitely vaccine related or study procedure related. Per protocol, the extension study included data from 9- to 15-year-old females regardless of lot administered.
Time Frame: Up to ~Month 126
Population: All participants who received at least 1 study vaccination in the base study and had follow-up data.
Measure: Number; unit: Percentage of Participants
Arm/Group | Extension Study: 9- to 15-Year-Old Females | Extension Study: 9- to 15-Year-Old Males
Number analyzed (Participants) | 971 | 301
Percentage of Participants | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: Base Study: Up to ~12 months; Extension Study: Up to ~126 months
Description: Base Study and Extension Study: ACM was analyzed in all randomized participants. Safety was analyzed in all participants who received at least one dose of 9vHPV and had available follow-up data, per protocol. ACM and safety were reported separately for base study, first extension (EXT1) and second extension (EXT2).
Groups:
- EXT1: 9- to 15-Year-Old Females; EXT1: 9- to 15-Year-Old Males: In the base study, participants received the 9vHPV L1 VLP vaccine (0.5 mL intramuscular injection) at Day 1, Month 2, and Month 6 and were evaluated through Month 12. In the extension study, the participants were followed up for safety and immunogenicity up to Month 36 (EXT1).
- EXT2: 9- to 15-Year-Old Females; EXT2: 9- to 15-Year-Old Males: In the base study, participants received the 9vHPV L1 VLP vaccine (0.5 mL intramuscular injection) at Day 1, Month 2, and Month 6 and were evaluated through Month 12. In the extension study, the participants were followed up for immunogenicity, effectiveness, and safety up to Month 126 (EXT2).
Arm/Group | Base Study: 9- to 15-Year-Old Females (Lot 1) | Base Study: 9- to 15-Year-Old Females (Lot 2) | Base Study: 9- to 15-Year-Old Females (Lot 3) | Base Study: 9- to 15-Year-Old Males (Lot 1) | Base Study: 16- to 26-Year-Old Females (Lot 1) | EXT1: 9- to 15-Year-Old Females | EXT1: 9- to 15-Year-Old Males | EXT2: 9- to 15-Year-Old Females | EXT2: 9- to 15-Year-Old Males
All-Cause Mortality (participants affected / at risk) | 0/648 | 0/643 | 0/644 | 0/669 | 0/470 | 1/1604 | 0/568 | 1/971 | 0/301
Serious Adverse Events (participants affected / at risk) | 6/643 | 2/639 | 8/641 | 11/662 | 15/466 | 2/1604 | 0/568 | 3/971 | 0/301
Other Adverse Events (participants affected / at risk) | 538/643 | 537/639 | 554/641 | 505/662 | 404/466 | 0/1604 | 0/568 | 0/971 | 0/301
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Base Study: 9- to 15-Year-Old Females (Lot 1) (N=643) | Base Study: 9- to 15-Year-Old Females (Lot 2) (N=639) | Base Study: 9- to 15-Year-Old Females (Lot 3) (N=641) | Base Study: 9- to 15-Year-Old Males (Lot 1) (N=662) | Base Study: 16- to 26-Year-Old Females (Lot 1) (N=466) | EXT1: 9- to 15-Year-Old Females (N=1604) | EXT1: 9- to 15-Year-Old Males (N=568) | EXT2: 9- to 15-Year-Old Females (N=971) | EXT2: 9- to 15-Year-Old Males (N=301)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disseminated tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain injury (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cervical incompetence (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Acute psychosis (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion induced (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Base Study: 9- to 15-Year-Old Females (Lot 1) (N=643) | Base Study: 9- to 15-Year-Old Females (Lot 2) (N=639) | Base Study: 9- to 15-Year-Old Females (Lot 3) (N=641) | Base Study: 9- to 15-Year-Old Males (Lot 1) (N=662) | Base Study: 16- to 26-Year-Old Females (Lot 1) (N=466) | EXT1: 9- to 15-Year-Old Females (N=1604) | EXT1: 9- to 15-Year-Old Males (N=568) | EXT2: 9- to 15-Year-Old Females (N=971) | EXT2: 9- to 15-Year-Old Males (N=301)
Injection site erythema (General disorders) | 184 (264) | 192 (287) | 195 (281) | 159 (219) | 132 (220) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 506 (1166) | 513 (1183) | 529 (1215) | 465 (919) | 393 (970) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 207 (317) | 237 (372) | 226 (380) | 173 (249) | 150 (261) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 76 (91) | 57 (67) | 64 (74) | 84 (94) | 43 (53) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 120 (182) | 122 (170) | 113 (156) | 98 (143) | 106 (166) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication guidelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-09-06): https://cdn.clinicaltrials.gov/large-docs/22/NCT00943722/Prot_SAP_000.pdf